CLINICAL TRIAL: NCT00913705
Title: Randomized Trial of Surgery With or Without Paclitaxel Plus Carboplatin as Neoadjuvant or Adjuvant Chemotherapy in Patients With Operable, Non-small-cell Lung Cancer
Brief Title: Neoadjuvant or Adjuvant Chemotherapy in Patients With Operable Non-small-cell Lung Cancer
Acronym: NATCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NATCH - GECP 99/02
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: NATCH; LUNG; OPERABLE NSCLC; SURGERY PLUS ADJUVANT THERAPY; SURGERY PLUS NEOADJUVANT THERAPY
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Neoadjuvant Therapy; Paclitaxel; Carboplatin; Chemotherapy, Adjuvant; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): The patients will be randomized to receive taxol (Paclitaxel) and carboplatin as adjuvant or as neoadjuvant regimen or to surgery alone
  Interventions: Drug: Neoadjuvant chemotherapy (taxol and carboplatin); Drug: Adjuvant chemotherapy (taxol and carboplatin); Procedure: Surgery

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy (taxol and carboplatin) — Taxol: 200mg/m2 infusion over 3 hours; Carboplatin: AUC= 6 at the end of the Taxol infusion. Administration of 3 cycles at 21-day intervals. Prior to surgery.
Drug: Adjuvant chemotherapy (taxol and carboplatin) — Taxol: 200mg/m2 infusion over 3 hours; Carboplatin: AUC= 6 at the end of the Taxol infusion. Administration of 3 cycles at 21 days interval. Post-surgery
Procedure: Surgery — Surgery

SUMMARY:
Open-label multicenter randomized Phase III trial.

DETAILED DESCRIPTION:
Randomized trial of surgery with or without Paclitaxel (taxol) plus Carboplatin as neoadjuvant or adjuvant chemotherapy in patients with operable, non-small-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patients eligible for the study are those with a diagnosis, histologically or cytologically proven, of NSCLC without metastases at stages IB, IIA, IIB and IIIA (not N2) of the disease. Patients with stage IA and tumor size >2cm will be eligible as well.
* Patients aged > 18 years.
* Tumor considered resectable by the attending surgeon.
* The patient must have an ECOG *2 or Karnofsky >60%.
* The patients need to have adequate hematological, renal and hepatic function defined as:

Absolute neutrophil counts (ANC*) *1.5 x 109/L Platelet counts *100 x 109/L Total bilirubin *1.25 x upper limit of normal distribution Serum creatinine <120 umol/L (<1.5 mg/dl) Creatinine clearance >60 ml/min

* ANC = segmented neutrophils + banded neutrophils

  * The patients should have recovered from any serious surgical sequellae.
  * Informed consent must be obtained from the patient in accordance with the requirements of the IRB/EC.
  * If female, the patient must not be pregnant or breast-feeding. Women of child bearing potential need to have a pregnancy test performed and to take appropriate contraceptive action during the period of the study.
  * Operability criteria: Lung function test will be performed so as to confirm a predictive postoperative value of FEV-1 >-800 ml, i.e. correct homeostasis. A carbon monoxide diffusion test is to be conducted and, when applicable, repeated following the induction treatment while taking into account the sensitivity of post-chemotherapy pulmonary toxicity detection.

Exclusion Criteria:

* Patients who have previously been treated with chemotherapy and/or radiotherapy.
* History of significant cardiovascular disease such as non-controlled hypertension, unstable angina or congestive heart failure even if these are controlled by medication. Documented history of acute myocardial infarction in the previous year, ventricular arrhythmias that required medication or 2nd or 3rd atrial-ventricular blocks.
* Pre-existing sensory or motor neurotoxicity grade >2 based on the WHO criteria.
* Active infection or other clinical state that could seriously reduce the patient's capacity to tolerate the treatment protocol, including previous allergic reactions to products containing Cremophor (e.g. cyclosporin or vitamin K).
* Previous or concomitant malignant tumor (with the exception of in situ cervical carcinoma, baso-cellular carcinoma, squamous cell skin carcinoma or urothelial superficial carcinoma) which are considered potentially curable with oncological treatment and have a disease free survival (DFS) greater than 5 years EXCEPTING breast cancer, melanoma and hypernephroma
* Marked psychoses or senility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Estimated)
Dates: Start 1999-09; Primary Completion 2007-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Evaluate disease-free survival (DFS) and overall survival (OS) | 5 years
  DFS: defined as the length of time from the date of diagnosis to the date of the first documented progression of disease OS: defined as the length of time from either the date of diagnosis or the start of the treatment that patients diagnosed with the disease are still alive.

SECONDARY OUTCOMES:
Evaluate levels of response and the adverse effects of the chemotherapy | 5 years
  Occurrence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Enriqueta Felip, MD, Principal Investigator — HOSPITAL VALL D'HEBRON (Barcelona); Rafael Rosell, MD, Principal Investigator — ICO-HOSPITAL UNIV. GERMANS TRIAS I PUJOL (Badalona)

REFERENCES:
- [Result] Felip E, Rosell R, Maestre JA, Rodriguez-Paniagua JM, Moran T, Astudillo J, Alonso G, Borro JM, Gonzalez-Larriba JL, Torres A, Camps C, Guijarro R, Isla D, Aguilo R, Alberola V, Padilla J, Sanchez-Palencia A, Sanchez JJ, Hermosilla E, Massuti B; Spanish Lung Cancer Group. Preoperative chemotherapy plus surgery versus surgery plus adjuvant chemotherapy versus surgery alone in early-stage non-small-cell lung cancer. J Clin Oncol. 2010 Jul 1;28(19):3138-45. doi: 10.1200/JCO.2009.27.6204. Epub 2010 Jun 1. PMID 20516435
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org